CLINICAL TRIAL: NCT07352098
Title: Efficacy and Safety of Short-Term, High-Dose Vonoprazan-Based Dual Therapy Versus Standard-Dose Vonoprazan-Based Dual Therapy for Helicobacter Pylori Eradication: A Multicenter, Open-Label, Randomized Controlled Trial
Brief Title: 7-day High-Dose Vonoprazan-amoxicillin Dual Therapy Versus 14-day Vonoprazan-amoxicillin Dual Therapy for H. Pylori
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yueyue Li (Other)
Collaborators: Qilu Hospital of Shandong University (Other); Shandong University of Traditional Chinese Medicine (Other); Zaozhuang Municipal Hospital (Other); Qilu Hospital of Shandong University, Dezhou Branch (Unknown); Yantai Zhifu Hospital (Unknown); Kashi Prefecture Hospital of Traditional Chinese Medicine (Unknown); Guanxian People's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Yueyue Li, associate chief physician, Qilu Hospital of Shandong University
Organization: Qilu Hospital of Shandong University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202510
Record Dates: First submitted 2026-01-07; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Helicobacter
Keywords: dual therapy; short term

STUDY DESIGN:
Intervention Model Description: Participants with Helicobacter pylori infection will be randomly assigned in a 1:1 ratio to one of two treatment groups:
  * A 7-day high-dose vonoprazan-amoxicillin dual therapy group: vonoprazan 20 mg three times daily + amoxicillin 1,000 mg three times daily, administered orally for 7 days.
  * A 14-day vonoprazan-amoxicillin dual therapy group: vonoprazan 20 mg twice daily + amoxicillin 1,000 mg three times daily, administered orally for 14 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 7-day high-dose vonoprazan-amoxicillin dual therapy group (Experimental)
  Interventions: Drug: 7-day high-dose vonoprazan-amoxicillin dual therapy group
- 14-day vonoprazan-amoxicillin dual therapy group (Experimental)
  Interventions: Drug: 14-day vonoprazan-amoxicillin dual therapy group

INTERVENTIONS:
Drug: 7-day high-dose vonoprazan-amoxicillin dual therapy group — Patients in the 7-day high-dose vonoprazan-amoxicillin dual therapy group received vonoprazan fumarate tablets 20 mg three times daily, administered 30 minutes before meals, and amoxicillin 1,000 mg three times daily, taken after meals.
  Both medications were administered orally for 7 consecutive days.
  Arms: 7-day high-dose vonoprazan-amoxicillin dual therapy group
Drug: 14-day vonoprazan-amoxicillin dual therapy group — Patients in the 14-day vonoprazan-amoxicillin dual therapy group received vonoprazan fumarate tablets 20 mg twice daily, administered 30 minutes before meals, and amoxicillin 1,000 mg three times daily, taken after meals.
  Both medications were administered orally for 14 consecutive days.
  Arms: 14-day vonoprazan-amoxicillin dual therapy group

SUMMARY:
Helicobacter pylori infection is a prevalent global gastrointestinal condition linked to chronic gastritis, peptic ulcer disease, and gastric cancer. Potent and sustained acid suppression improves eradication efficacy. Vonoprazan, a potassium-competitive acid blocker, provides rapid and stable acid inhibition and has become an important component of dual therapy with amoxicillin. However, the optimal dosing strategy and treatment duration for vonoprazan-based dual therapy are not yet fully established.

This multicenter, open-label, randomized controlled trial compares the efficacy and safety of a short-term, high-dose vonoprazan-based dual therapy (20 mg three times daily for 7 days) with a standard-dose regimen (20 mg twice daily for 14 days), both combined with amoxicillin, for first-line H. pylori eradication. Adult participants with confirmed H. pylori infection will be randomized 1:1 to the two treatment groups. The primary outcome is the eradication rate of H. pylori at 6 weeks after completion of therapy. Secondary outcomes include safety assessments and medication adherence. This study will provide evidence on whether a higher dose and shorter treatment course can achieve similar eradication rates with acceptable safety and tolerability compared to the standard regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years, no gender restrictions;
* Patients with H. pylori infection confirmed by 13C/14C-urea breath test ;
* No prior history of H. pylori eradication therapy;

Exclusion Criteria:

* Patients allergic to study medications (vonoprazan fumarate, amoxicillin);
* Patients with active qastrointestinal bleeding,;
* Patients undergone or scheduled to undergo surgery within 1 month prior to randomization or during the study period that may affect gastric acid secretion (e.g., gastric surgery, vagotomy, or craniotomy);
* Patients underlying severe medical conditions deemed by the investigator to potentially confound study results or compromise subject safety, such as: hepatic impairment (ALT or AST > 1.5 times the upper limit of normal); renal impairment (Cr ≥ 2.0 mg/dL or eGFR < 50 mL/min/1.73 m²); immunosuppression; malignancy; severe central nervous system, cardiovascular, or respiratory disease;
* Patients with medication history of bismuth, antibiotics within 4 weeks, or proton pump inhibitors within 2 weeks;
* Patients with behaviors potentially increasing disease risk: history of chronic substance abuse or alcohol dependence within 12 months prior to screening;
* Patients planning pregnancy, currently pregnant, breastfeeding, or unwilling to use contraception during the trial period;
* Patients unable or unwilling to provide informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | 6 weeks after treatment

SECONDARY OUTCOMES:
incidence of adverse events | immediately after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Kashi Prefecture Hospital of Traditional Chinese Medicine, Kashgar, Xinjiang, China

IPD SHARING:
Plan to Share IPD: No